CLINICAL TRIAL: NCT00765466
Title: A Phase II Open Label, Multi-Center Study With AVR118 in Anorectic Patients With Recurrent or Advanced Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study transferred out of McGill because PI relocted to another insitution.
Sponsor: McGill University (Other)
Responsible Party: Dr. Martin Chasen, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McG 0710
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2007-03

CONDITIONS: Cancer
Keywords: Explore the effect of AVR118 4.0 mL, given subcutaneously on appetite
MeSH Terms: conditions — Neoplasms | interventions — EOM613

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AVR118 — daily doses of 4.0 mL AVR118 subcutaneously

SUMMARY:
This is an open label, Phase II, multi-center study designed to evaluate the effect of AVR118 when administered to patients with systemic symptoms related to recurrent or metastatic cancers who may or may not be undergoing anti-cancer treatment. During the initial, induction treatment phase of the study, AVR118, 4.0 mL, will be given subcutaneously each day for 28 days. Patients who respond to the trial period dosing will be eligible to continue on AVR118 if they and their physicians believe it would be beneficial, and if no safety concerns are raised.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor cancer, leukemia, lymphoma, or multiple myeloma.
* Concurrent anti-cancer treatment, such as chemotherapy or radiation therapy is permitted except for neo-adjuvant or adjuvant programs.
* Between the ages of 18-85.
* Symptoms of recurrent or metastatic cancer in which anorexia is a predominant symptom, not necessarily associated with cachexia, and are not attributed to anemia, concomitant illnesses, or obstruction or loss of organ function.
* Karnofsky performance status of 40%
* Palliative Prognostic Score (PaP) of less than 6
* Patient is expected to be able to remain on a study protocol for two months.
* Pretreatment laboratory data within 7 days of enrollment:
* Hemoglobin >8.5 g/dL , or on stable doses (hematocrit stable within 1 gram and dose stable for one month) of erythropoietin or similar medication.
* Absolute neutrophil count (ANC) 1,500/mm3.
* Platelets 50,000/mm3.
* Total bilirubin 2.0
* ALT and AST 2.5 times the ULN, or, if the patient has liver metastases, 5 times the ULN.
* Creatinine 1.5 mg/dL.
* Normal TSH
* Testosterone levels determined.
* Voluntary written informed consent before performance of any study-related procedure that is not part of normal medical care.
* Ability to self-administer subcutaneous medication if an assistant or nurse is not available, and to keep a compliance journal documenting injections at home.
* If on an antidepressant, the dose must have been stabilized for at least 30 days.
* Female patient is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable barrier method for contraception during the study

Exclusion Criteria:

* Patient has uncontrolled brain metastases or central nervous system disease.
* Patient has mechanical, non-reversible reason for not being able to eat, or have a potential for developing malignant bowel obstruction during the course of the induction phase of treatment, or patients requiring a PEG for obstruction.
* Patient has had any major surgery within four weeks of enrollment.
* Patient has an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* In the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Female patient is pregnant or breast-feeding.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Karnofsky Performance Status Disease-related symptoms: ESAS and PG-SGA Anorexia Weight Lean Body Mass, Triceps skin fold, and grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Maribel de Diego, Ph.D., Study Director — Advances Viral Research Corporation
Locations (1):
- McGill University Clinical Research Program, Montreal, Quebec, Canada